CLINICAL TRIAL: NCT03726502
Title: Comparing Uretersocopy With Versus Without Use of Guide-wire in Treatment of Ureteral Stone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Shemshaki, Director, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Q12133
Record Dates: First submitted 2017-04-19; First posted 2018-10-31 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-10

CONDITIONS: Ureteral Calculi
Keywords: Ureteral Calculi; safety guide-wire; ureteroscopy
MeSH Terms: conditions — Ureteral Calculi | interventions — Ureteroscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ureteroscopy with safety guide-wire (Active Comparator): ureteroscopy is done with use of safety guide-wire, this is a one procedure that we use safety guide wire (as a device) during ureteroscopy
  Interventions: Procedure: ureteroscopy with safety guide-wire; Procedure: with safety guide-wire
- ureteroscopy alone (Placebo Comparator): ureteroscopy is done without use of safety guide-wire, this is a one procedure that we don"t use safety guide wire (as a device) during ureteroscopy
  Interventions: Procedure: ureteroscopy alone; Procedure: without safety guide-wire
- with safety guide-wire (Active Comparator): ureteroscopy is done with use of safety guide-wire, this is a one procedure that we use safety guide wire (as a device) during ureteroscopy
  Interventions: Procedure: ureteroscopy with safety guide-wire; Procedure: with safety guide-wire
- without safety guide-wire (Placebo Comparator): ureteroscopy is done without use of safety guide-wire, this is a one procedure that we don"t use safety guide wire (as a device) during ureteroscopy
  Interventions: Procedure: ureteroscopy alone; Procedure: without safety guide-wire

INTERVENTIONS:
Procedure: ureteroscopy with safety guide-wire — ureteroscopy with use of safety guide-wire in treatment of ureteral stone
  Arms: ureteroscopy with safety guide-wire; with safety guide-wire
Procedure: ureteroscopy alone — ureteroscopy without use of safety guide-wire in treatment of ureteral stone
  Arms: ureteroscopy alone; without safety guide-wire
Procedure: without safety guide-wire — ureteroscopy without use of safety guide-wire in treatment of ureteral stone
  Arms: ureteroscopy alone; without safety guide-wire
Procedure: with safety guide-wire — ureteroscopy with use of safety guide-wire in treatment of ureteral stone
  Arms: ureteroscopy with safety guide-wire; with safety guide-wire

SUMMARY:
The purpose of this study is to compare ureteroscopy with and without use of safety guide-wire in treatment of ureteral stone

DETAILED DESCRIPTION:
While there are some retrospective studies compared ureteroscopy with and without use of safety guide-wire in treatment of ureteral stone, there is not randomized clinical trial in this regard. This study was designed to compare the efficacy and safety of ureteroscopy with and without use of safety guide-wire in treatment of ureteral stone

ELIGIBILITY:
Inclusion Criteria:

* ureteral stone who underwent ureteroscopy

Exclusion Criteria:

* transplant kidney
* coagulopathy disorders
* history of ureteral stenosis
* skeletal disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
stone free rate | 3 months after surgery
  rate of patients without any residue of stone

SECONDARY OUTCOMES:
operation time | at time of surgery
  the time between insertion of ureteroscopy till insertion of catheter
grade of kidney hydronephrosis | 3 months after surgery
  grade of hydronephrosis is classified as: 0-4 grades
ureteral injury | at time of surgery
  ureteral injury is classified as: Mucosal abrasion, Ureteral perforation, Intussusception / avulsion

CONTACTS AND LOCATIONS:
Overall Officials: Abbas Basiri, prof, Study Chair — Shahid beheshty university of medical sciences
Locations (1):
- Shahid beheshty university of medical sciences, Tehrān, Iran

IPD SHARING:
Plan to Share IPD: Undecided